CLINICAL TRIAL: NCT07033936
Title: Prevalence Of Irritable Bowel Syndrome, Its Risk Factors, And Impact On Increasing Anxiety And Depression Among Egyptian Medical Students
Brief Title: Prevalence of Irritable Bowel Syndrome Among Egyptian Medical Students
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZU-IRB # 1404/3-June-2025
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — An online Questionnaire will be shared via social media such as WhatsApp, Facebook or X for Egyptian medical students and intern to fill

SUMMARY:
Assess prevalence of irritable bowel syndrome among both medical students and medical interns, and the most significant risk factors of this condition, and highlight the association between IBS symptoms, anxiety & depression.

DETAILED DESCRIPTION:
One of the most common gastrointestinal disorders is irritable bowel syndrome (IBS). It is a chronic functional bowel disease in which abnormal bowel habits, such as diarrhea, constipation, or both, are associated with abdominal pain and distension. Around 11% of the general population suffers from their symptoms regardless of the geographical distribution.

Irritable bowel syndrome is more common among females and patients younger than 50. For medical students, IBS is common and may affect up to 25% of them.. Especially final-year students, due to the increasing workload of the final year.

Several risk factors increase the prevalence of irritable bowel syndrome, including environmental factors, life events, and junk food abuse. Also, Psychological disorders as severe levels of anxiety, depression, and stress, may contribute to the occurrence of irritable bowel syndrome, and this can be explained by the pathophysiology of IBS, maybe by brain-gut interaction.

Globally, the prevalence of anxiety and depression is higher in medical students compared to other populations, as it reaches up to 38.7% among them. Many factors play a role in increasing the prevalence of anxiety and depression among medical students as stressful courses in medical study, exposure to the death of patients, and others. In Egypt, the prevalence of medical students suffering from stress and anxiety is high due to several problems as financial problems, work overload, traditional methods of education, and the increasing number of students, making communication with thePage 3 of 9 lecturer difficult and that increase incidence of IBS among Egyptian medical students.

Just as anxiety is considered a risk factor for the development of Irritable Bowel Syndrome (IBS), IBS can also lead to the occurrence of anxiety and depression, and that can be explained by brain-gut interaction.

Patients with IBS have a three-times increased risk of either anxiety or depression, compared to healthy subjects.

Although the importance of this topic is recognized, there are limited data about the exact prevalence of irritable bowel syndrome among medical students in Egypt.

Previous studies have discussed this topic in three medical schools in Egypt, but their sample size were too small, and they did not assess the associated anxiety and depression among these students, so no definitive conclusion can be made. This is the first study in Zagazig University hospital to assess the prevalence of irritable bowel syndrome among both medical students and medical interns, and the most significant risk factors of this condition, and highlight the association between IBS symptoms and anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian Medical students and interns
* Their age ranges from 18 to 29 years
* Have access to online platforms such as Facebook, WhatsApp, and Telegram.
* Accept to participate in the questionnaire

Exclusion Criteria:

* Participate who refused to participate

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian Medical students and Intern
Sampling Method: Non-Probability Sample
Enrollment: 1093 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-06 (Actual)

PRIMARY OUTCOMES:
Number of irritable bowel syndrome patients among population | 1 month
  Will use Rome IV criteria to diagnose IBS. It is composed of three questions about the presence of GIT symptoms. The presence of at least two of the three diagnoses the IBS.

SECONDARY OUTCOMES:
Number of IBS patients suffering anxiety and depression | 1 month
  Will use the HAD questionnaire to diagnose both anxiety and depression. It is a 14 questionnaire divided into two subscales, one for anxiety and the other for depression. Each question is composed of 4 answers, scored from 0 to 3. Cumulative score for each subscale determines the level of either anxiety or depression. an individual can score between 0 and 21 for either anxiety or depression, and be classified into the following categories: 0 to 7, normal; 8 to 10, borderline; and 11 to 21, abnormal (case)

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Faculty of Medicine and Affiliated Hospital, Zagazig, Egypt

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820

DOCUMENTS (1):
  • Study Protocol (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT07033936/Prot_001.pdf